CLINICAL TRIAL: NCT01095224
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Heterologous Prime-Boost Regimens Utilizing Recombinant Adenovirus Serotype 35 (rAd35) With HIV-1 Clade A Env Insert and Recombinant Adenovirus Serotype 5 (rAd5) With HIV-1 Clade A or B Env Inserts in Healthy, HIV-1-Uninfected Adults
Brief Title: Evaluating Heterologous-Insert Prime-Boost HIV Vaccine Regimens in HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 083; 10783 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- rAd35 Env A and rAd5 Env A (Experimental): Participants will receive the rAd35 Env A vaccine at baseline and the rAd5 Env A vaccine at Month 3.
  Interventions: Biological: rAd35 Env A; Biological: rAd5 Env A
- rAd35 Env A and rAd5 Env B (Experimental): Participants will receive the rAd35 Env A vaccine at baseline and the rAd5 Env B vaccine at Month 3.
  Interventions: Biological: rAd35 Env A; Biological: rAd5 Env B
- rAd35 Env A and rAd35 Env A (Experimental): Participants will receive the rAd35 Env A vaccine at baseline and at Month 3.
  Interventions: Biological: rAd35 Env A
- rAd5 Env A and rAd5 Env A (Experimental): Participants will receive the rAd5 Env A vaccine at baseline and at Month 3.
  Interventions: Biological: rAd5 Env A
- rAd5 Env A and rAd5 Env B (Experimental): Participants will receive the rAd5 Env A vaccine at baseline and the rAd5 Env B vaccine at Month 3.
  Interventions: Biological: rAd5 Env A; Biological: rAd5 Env B

INTERVENTIONS:
Biological: rAd35 Env A — 1 x 10^10 particle units (PU) administered as 1 mL intramuscularly (IM) in deltoid
  Other Names: VRC-HIVADV027-00-VP
  Arms: rAd35 Env A and rAd35 Env A; rAd35 Env A and rAd5 Env A; rAd35 Env A and rAd5 Env B
Biological: rAd5 Env A — 1 x 10^10 PU administered as 1 mL IM in deltoid
  Other Names: VRC-HIVADV038-00-VP
  Arms: rAd35 Env A and rAd5 Env A; rAd5 Env A and rAd5 Env A; rAd5 Env A and rAd5 Env B
Biological: rAd5 Env B — 1 x 10^10 PU administered as 1 mL IM in deltoid
  Other Names: VRC-HIVADV052-00-VP
  Arms: rAd35 Env A and rAd5 Env B; rAd5 Env A and rAd5 Env B

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of an adenovirus-based HIV-1 vaccine regimen that includes two vaccines given at different time points in HIV-uninfected adults.

DETAILED DESCRIPTION:
One approach to developing a preventive HIV vaccine includes the use of a prime-boost vaccine strategy. This type of strategy involves two vaccines, given sequentially at different time points. The goal is to stimulate different parts of the immune system and enhance the body's overall immune response to HIV. In this study, participants will receive two HIV vaccines 3 months apart. Heterologous-insert prime-boost vaccine regimens, which use the same gene from different HIV-1 subtypes, may be more effective than traditional homologous insert prime-boost vaccine regimens at eliciting immune responses directed at epitopes that are highly prevalent, possibly leading to a more effective immune system response to the vaccine. The purpose of this study is to assess the safety and immunogenicity of a heterologous-insert prime-boost HIV vaccine regimen that uses inserts from different HIV-1 subtypes and different adenovirus vectors.

This study will enroll healthy, HIV-uninfected people. Participants will be randomly assigned to one of five study groups:

* Group 1 will receive the recombinant adenovirus serotype 35 (rAd35) Env A vaccine at baseline and the recombinant adenovirus serotype 5 (rAd5) Env A vaccine at Month 3.
* Group 2 will receive the rAd35 Env A vaccine at baseline and the rAd5 Env B vaccine at Month 3.
* Group 3 will receive the rAd35 Env A vaccine at baseline and at Month 3.
* Group 4 will receive the rAd5 Env A vaccine at baseline and at Month 3.
* Group 5 will receive the rAd5 Env A vaccine at baseline and the rAd5 Env B vaccine at Month 3.

All vaccines will be injected into the upper arm. At both vaccination study visits, participants will undergo a physical exam, a medical and medication history review, a blood and urine collection, and questionnaires. Participants will receive counseling on HIV risk reduction and pregnancy prevention. After receiving the vaccine, participants will remain in the clinic for at least 30 minutes for observation and monitoring of side effects. For 3 days after each vaccination, participants will record their temperature and side effects in a symptom log. In addition to the vaccine study visits, other study visits will occur at Week 2, two weeks after the Month 3 visit, and at Months 4, 6, and 9, at which time various study procedures will be repeated.

Participants will be contacted by study researchers once a year for 5 years for follow-up safety monitoring. Safety monitoring will not involve visiting a clinic except if a confirmatory HIV test is needed. Questions will assess health and adverse events.

The primary objective of this study is to assess the safety and tolerability, as well as the ability, of a heterologous-insert prime-boost vaccine regimen using env inserts from different HIV-1 clades to increase T-cell responses. In addition, this study is evaluating the effectiveness of a heterologous-insert prime-boost and vector prime-boost vaccine regimen at increasing T-cell responses. The study will also compare the degree of polyfunctionality of insert specific T cells after vaccination within heterologous and homologous vector vaccine regimens.

ELIGIBILITY:
Inclusion Criteria:

* Assessed by clinic staff as being "low risk" for HIV infection
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willing to be followed for the duration of the study
* Able and willing to provide informed consent
* Assessment of understanding, including the completion of a questionnaire before the first vaccination and demonstration of understanding for all questionnaire items answered incorrectly
* Willing to receive HIV test results
* Willing to discuss HIV infection risks, amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required study visit
* Willing to continue annual follow-up contact after the final study visit for a total of 5 years after study entry
* In good general health, as shown by medical history, physical exam, and screening laboratory tests
* Assessed by the clinic staff as having a low risk of HIV infection on the basis of sexual behaviors in the 12 months before study entry. More information on this criterion can be found in the protocol.
* Adenovirus 5 nAb titer less than 1:18
* Adenovirus 35 nAb titer less than 1:12
* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female and greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell (WBC) count between 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within site's normal range or with site physician approval
* Platelet level between 125,000 to 550,000/mm^3
* Alanine aminotransferase (ALT) less than or equal to 1.25 times the site's upper limit of normal
* Negative HIV-1 and -2 blood test
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV test is positive
* Normal urine test results
* Participants who were born female must have a negative pregnancy test result before the first study vaccination
* Participants who were born female must agree to use an effective form of contraception from at least 21 days before study entry until the last study visit. More information on this criterion can be found in the protocol.
* Participants who were born female must agree not to seek pregnancy through alternative methods (e.g., artificial insemination, in vitro fertilization) until after the last study visit
* If born male, must be fully circumcised (as documented at screening examination)

Exclusion Criteria:

* Excessive daily alcohol use, frequent binge drinking, chronic marijuana abuse, or use of any other illicit drugs in the 12 months before study entry
* History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B in the 12 months before study entry
* Received non-HIV experimental vaccines in a previous vaccine trial in the 5 years before study entry
* Received HIV vaccines in a prior HIV vaccine trial
* Immunosuppressive medications received within 168 days before the first study vaccination
* Blood products received within 120 days before the first study vaccination
* Immunoglobulin received within 60 days before the first study vaccination
* Live attenuated vaccines received within 30 days before the first study vaccination or scheduled within 14 days after injection
* Investigational research agents received within 30 days before the first study vaccination
* Intent to participate in another investigational drug study
* Any vaccines that are not live attenuated vaccines and were received within 14 days before the first study vaccination
* Allergy treatment with antigen injections within 30 days before the first study vaccination or scheduled within 14 days after the first vaccination
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, abnormal physical examination findings, clinically significant abnormal laboratory results, or past medical history that may affect current health
* Any medical, psychiatric, occupational, or other condition that would interfere with participation in the study
* Serious adverse reactions to vaccines, including anaphylaxis and related symptoms (e.g., hives, respiratory difficulty, angioedema, abdominal pain). A person who had an adverse reaction to the pertussis vaccine is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection
* Asthma, other than mild well-controlled asthma. More information on this criterion can be found in the protocol.
* Type 1 or type 2 diabetes mellitus, including cases controlled with diet alone. People with a history of gestational diabetes are not excluded.
* Surgical removal of the thyroid or thyroid disease requiring medication in the 12 months before study entry
* Angioedema in the 3 years before study entry or angioedema requiring medication in the 2 years before study entry
* High blood pressure that is not well controlled or high blood pressure of 150/100 mm Hg or greater at study entry. More information on this criterion can be found in the protocol.
* Body mass index (BMI) greater than or equal to 40, or BMI greater than or equal to 35 and two or more of the following conditions: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia
* Bleeding disorder (e.g., factor deficiency, coagulopathy, platelet disorder requiring special precautions)
* Cancer. People with surgically removed cancer, that in the opinion of the investigator, is unlikely to recur during the study period are not excluded.
* Seizure disorder. People with a history of seizures who have not required medications or had a seizure within the 3 years before study entry are not excluded.
* Absence of the spleen
* Psychiatric condition that makes study compliance difficult (e.g., people with psychoses in the 3 years before study entry, ongoing risk for suicide, history of suicide attempt in the 3 years before study entry)
* Pregnant or breastfeeding
* Has been circumcised within 90 days prior to first vaccination or displays evidence that surgical site is not fully healed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local injection site reactogenicity signs and symptoms, including pain, tenderness, erythema, induration, and maximum severity of pain and/or tenderness | Measured at baseline and Month 3
Frequency and severity of systemic reactogenicity signs and symptoms, including fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and maximum severity of systemic symptoms | Measured at baseline and Month 3
Frequency of adverse events (AEs) categorized by MedDRA body system, MedDRA preferred term, severity and assessed relationship to study products; detailed description of all AEs meeting DAIDS criteria for expedited reporting | Measured at Month 9
Distribution of values of safety laboratory measures, including white blood cells (WBCs), neutrophils, lymphocytes, hemoglobin, platelets, and alanine aminotransferase (ALT) at baseline and at postvaccination follow-up study visits | Measured at Month 9
Number of participants with early discontinuation of vaccinations and reason for discontinuation | Measured at Month 9
Number of shared HIV epitopes targeted by T-cells | Measured at 4 weeks following the final vaccination
HIV-1-specific interferon gamma (IFN-y) ELISpot responses | Measured at 4 weeks following the final vaccination

SECONDARY OUTCOMES:
Number of shared HIV epitopes targeted by T-cells | Measured at 4 weeks following the final vaccination
HIV-1-specific IFN-y ELISpot responses | Measured at 4 weeks following the final vaccination
Frequency of insert-specific CD4 and CD8 cells | Measured at 4 weeks following the final vaccination
Number of HIV epitopes targeted by T-cells | Measured at 4 weeks following the final vaccination
Functional spectrum of CD4 and CD8 cells by intracellular cytokine staining (ICS) assay for IFN-y, IL-2, and TNF-a | Measured at Month 9
Binding and neutralizing antibody titers | Measured at baseline and at 4 weeks following the final vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Xia Jin, MD, PhD, Study Chair — University of Rochester
Locations (8):
- United States (8):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee

REFERENCES:
- [Background] Vaine M, Lu S, Wang S. Progress on the induction of neutralizing antibodies against HIV type 1 (HIV-1). BioDrugs. 2009;23(3):137-53. doi: 10.2165/00063030-200923030-00001. PMID 19627166
- [Background] Appay V, Douek DC, Price DA. CD8+ T cell efficacy in vaccination and disease. Nat Med. 2008 Jun;14(6):623-8. doi: 10.1038/nm.f.1774. PMID 18535580
- [Derived] Walsh SR, Moodie Z, Fiore-Gartland AJ, Morgan C, Wilck MB, Hammer SM, Buchbinder SP, Kalams SA, Goepfert PA, Mulligan MJ, Keefer MC, Baden LR, Swann EM, Grant S, Ahmed H, Li F, Hertz T, Self SG, Friedrich D, Frahm N, Liao HX, Montefiori DC, Tomaras GD, McElrath MJ, Hural J, Graham BS, Jin X; HVTN 083 Study Group and the NIAID HVTN. Vaccination With Heterologous HIV-1 Envelope Sequences and Heterologous Adenovirus Vectors Increases T-Cell Responses to Conserved Regions: HVTN 083. J Infect Dis. 2016 Feb 15;213(4):541-50. doi: 10.1093/infdis/jiv496. Epub 2015 Oct 15. PMID 26475930